CLINICAL TRIAL: NCT06658340
Title: Positivity in Post-COVID: Promoting Well-being in Patients with Post-COVID-19 Syndrome - a Feasibility and Acceptability Study
Brief Title: Feasibility of a Well-being Promotion Self-management Intervention in Post-COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Twente (Other)
Responsible Party: Principal Investigator, Gerko Schaap, Principal investigator, University of Twente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 241040
Record Dates: First submitted 2024-10-16; First posted 2024-10-26 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Post-COVID-19 Syndrome
Keywords: mental well-being; positive psychological intervention; self-management; long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention: Positivity in Post-COVID (Experimental): Participants will go through the training using a workbook for 12 consecutive days, once a day for 10-15 minutes.
  Interventions: Behavioral: Positivity in Post-COVID

INTERVENTIONS:
Behavioral: Positivity in Post-COVID — A training to support well-being and self-management in patients with post-COVID-19 syndrome

SUMMARY:
A training comprised of positive psychological interventions set out to improve mental well-being was developed for post-COVID-19 patients. This study aims to evaluate the feasibility and acceptability of this training.

DETAILED DESCRIPTION:
Research has shown that the quality of life and well-being of post-COVID-19 patients are often reduced, and that many patients struggle with self-management tasks, such as symptom management and emotion regulation. Training in self-management skills related to positive emotions, such as positive affect savouring, might help with these and can be provided prior to or in parallel with usual treatment. This study aims to investigate whether a training to improve the mental well-being is feasible and acceptable for people with post-COVID-19 syndrome. The training to be provided is based on previously evaluated sets of positive psychological interventions ('This is your life' and 'Training in Positivity') and adapted to a post-COVID-19 population. As a secondary aim, preliminary effectiveness will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Strongly suspected or clinically confirmed post-COVID-19 syndrome, i.e. confirmed symptoms persisting for at least 3 months after strongly suspected or confirmed SARS-CoV-2 infection
* Ages ≥18 years
* Dutch proficiency
* Provided informed consent

Exclusion Criteria:

* Recent (<5 years) diagnosis of a mood disorder, anxiety disorder or other psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-07-14 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention exercises | At post-intervention (2 weeks after baseline)
  Feasibility is assessed using items asking how often exercises were executed (never, 1, 2 or 3 times).
Acceptability of the intervention exercises - willingness to do again | At post-intervention (2 weeks after baseline) and at follow-up (6 weeks after baseline). Interviews are to be conducted soon after the post-questionnaire
  Acceptability is assessed using items on willingness to do again, satisfaction, perceived utility, experienced ease-of-use, experienced discomfort, and willingness to recommend to a) other patients and b) friends. Each item is measured on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), and assessed on an item level.
Acceptability of the intervention exercises - satisfaction | At post-intervention (2 weeks after baseline) and at follow-up (6 weeks after baseline). Interviews are to be conducted soon after the post-questionnaire
  Acceptability is assessed using items on willingness to do again, satisfaction, perceived utility, experienced ease-of-use, experienced discomfort, and willingness to recommend to a) other patients and b) friends. Each item is measured on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), and assessed on an item level.
Acceptability of the intervention exercises - perceived utility | At post-intervention (2 weeks after baseline) and at follow-up (6 weeks after baseline). Interviews are to be conducted soon after the post-questionnaire
  Acceptability is assessed using items on willingness to do again, satisfaction, perceived utility, experienced ease-of-use, experienced discomfort, and willingness to recommend to a) other patients and b) friends. Each item is measured on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), and assessed on an item level.
Acceptability of the intervention exercises - experienced ease-of-use | At post-intervention (2 weeks after baseline)
  Acceptability is assessed using items on willingness to do again, satisfaction, perceived utility, experienced ease-of-use, experienced discomfort, and willingness to recommend to a) other patients and b) friends. Each item is measured on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), and assessed on an item level.
Acceptability of the intervention exercises - experienced discomfort | At post-intervention (2 weeks after baseline)
  Acceptability is assessed using items on willingness to do again, satisfaction, perceived utility, experienced ease-of-use, experienced discomfort, and willingness to recommend to a) other patients and b) friends. Each item is measured on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), and assessed on an item level.
Acceptability of the intervention exercises - willingness to recommend | At post-intervention (2 weeks after baseline)
  Acceptability is assessed using items on willingness to do again, satisfaction, perceived utility, experienced ease-of-use, experienced discomfort, and willingness to recommend to a) other patients and b) friends. Each item is measured on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), and assessed on an item level.
Acceptability of the intervention exercises - interviews | Between post-intervention (2 weeks after baseline) and at follow-up (6 weeks after baseline).
  Acceptability will be further explored via in-depth interviews (optional in addition to the post- and follow-up questionnaires) and assessed using thematic analysis

SECONDARY OUTCOMES:
Change in affect | Baseline to post-intervention (2 weeks after baseline) and follow-up (6 weeks after baseline)
  Measured with the 20-item Positive and Negative Affect Schedule (PANAS). Positive affect (10 items) and negative affect (10 items) are assessed on a scale from 1 (not at all) to 5 (extremely) and calculated as sum scores. Higher scores indicate larger levels of positive and negative affect.
Change in mental well-being | Baseline to post-intervention (2 weeks after baseline) and follow-up (6 weeks after baseline)
  Measured with the 14-item Mental Health Continuum short form (MHC-SF), which assesses three subscales (emotional well-being via 3 items; psychological well-being via six items; and social well-being via five items) and a total mental well-being scale. Mean scores range between 0 - 5, with higher scores indicating more well-being.
Change in post-COVID symptom severity and functionality | Baseline to follow-up (6 weeks after baseline)
  Measured with the modified COVID-19 Yorkshire Rehabilitation Scale (C19YRSm) resulting in four subscales: symptom severity (0 - 30; higher scores indicating higher severity); functional ability (0 - 15; higher scores indicating higher dysfunction); presence of other symptoms (0 - 25; higher scores indicating more symptoms); and self-reported general health (0 - 10; higher scores indicating better health).
Change in fatigue | Baseline to post-intervention (2 weeks after baseline) and follow-up (6 weeks after baseline)
  Measured with the 4-item Short Fatigue Questionnaire (SFQ), resulting in one sum score of 4 - 28. Higher scores indicate more severe fatigue with scores ≥18 signalling clinically severe fatigue.
Change in anxiety | Baseline to post-intervention (2 weeks after baseline) and follow-up (6 weeks after baseline)
  Measured with the 14-item Hospital Anxiety and Depression Scale (HADS), with one subscale (7 items) on anxiety and one subscale (7 items) on depression. Sum scores range between 0 - 21 with higher scores (>7) indicating higher severity.
Change in depression | Baseline to post-intervention (2 weeks after baseline) and follow-up (6 weeks after baseline)
  Measured with the 14-item Hospital Anxiety and Depression Scale (HADS), with one subscale (7 items) on anxiety and one subscale (7 items) on depression. Sum scores range between 0 - 21 with higher scores (>7) indicating higher severity.
Change in ability to adapt | Baseline to follow-up (6 weeks after baseline)
  Ability to adapt is measured with the 10-item Generic Sense of Ability of Adapt Scale (GSAAS), resulting in a mean score between 0 - 4; higher scores indicating better sense of adaptability.
Change in perceived illness control | Baseline to follow-up (6 weeks after baseline)
  Illness perceptions, including perceived illness control and perceived treatment control, are measured with the brief Illness Perception Questionnaire (IPQ-K). Items are scored on range from 0 - 10, for control items higher scores indicating better perceived control.
Perceived overall impact | Between post-intervention (2 weeks after baseline) and follow-up (6 weeks after baseline)
  Perceived impact of the intervention will be explored via in-depth interviews (optional in addition to the post- and follow-up questionnaires).

OTHER OUTCOMES:
Recommendations for the intervention exercises | Between post-intervention (2 weeks after baseline) and follow-up (6 weeks after baseline)
  Recommendations for future interventions or iterations, including strengths of the training and motivation to participate, will be explored via in-depth interviews (optional in addition to the post- and follow-up questionnaires).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Twente, Enschede, Netherlands

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request